CLINICAL TRIAL: NCT06993194
Title: Comparison Between the Effects of Haloperidol and Dexmedetomidine on Delirium and Agitation in Patients With a Traumatic Brain Injury Admitted to the Intensive Care Unit
Brief Title: Comparison of Haloperidol and Dexmedetomidine for Delirium and Agitation in ICU Patients With Traumatic Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed El-Sayed Abdelghany Nasef, Resident of Anaesthesia and Intensive Care, Faculty of Medicine, Benha University, Egypt, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-990-2025
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury; Delirium; Agitation
Keywords: Traumatic Brain Injury; Delirium Management; Agitation in Intensive Care; Haloperidol; Dexmedetomidine; Sedation in Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Delirium; Psychomotor Agitation | interventions — Haloperidol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to one of two parallel groups. One group will receive haloperidol and the other will receive dexmedetomidine. Each group will follow a predefined drug protocol without crossover between groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: This is a double-blind study in which both the participants and the outcome assessors are unaware of the group assignments. Blinding is maintained through coded drug administration and identical infusion procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haloperidol Group (Active Comparator): Participants in this arm will receive intravenous haloperidol at a dose of 2.5 milligrams every eight hours, infused over ten minutes, starting 48 hours after admission to the intensive care unit. The intervention will continue for up to seven days or until resolution of delirium or agitation, whichever comes first. Rescue sedation with intravenous midazolam (1 milligram) and fentanyl (50 micrograms) may be administered if needed. Clinical assessments will include monitoring of delirium using the Confusion Assessment Method for the Intensive Care Unit, level of agitation using the Richmond Agitation-Sedation Scale, and consciousness using the Glasgow Coma Scale.
  Interventions: Drug: Haloperidol
- Dexmedetomidine Group (Experimental): Participants in this arm will receive intravenous dexmedetomidine at a dose of 0.5 micrograms per kilogram by continuous infusion, starting 48 hours after admission to the intensive care unit. The intervention will be administered every other day for up to seven days or until resolution of delirium or agitation. Rescue sedation with intravenous midazolam (1 milligram) and fentanyl (50 micrograms) may be administered if needed. Clinical assessments will include monitoring of delirium using the Confusion Assessment Method for the Intensive Care Unit, level of agitation using the Richmond Agitation-Sedation Scale, and consciousness using the Glasgow Coma Scale.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Haloperidol — Haloperidol will be administered intravenously at a dose of 2.5 milligrams every eight hours over ten minutes. Treatment will begin 48 hours after admission to the intensive care unit and will continue for up to seven days or until delirium and agitation resolve. The need for additional sedation will be addressed with intravenous midazolam and fentanyl as required. The patient's clinical status will be monitored using standardized assessments including the Confusion Assessment Method for the Intensive Care Unit and the Richmond Agitation-Sedation Scale.
  Arms: Haloperidol Group
Drug: Dexmedetomidine — Dexmedetomidine will be administered by continuous intravenous infusion at a dose of 0.5 micrograms per kilogram. Treatment will begin 48 hours after admission to the intensive care unit and will be repeated every other day for up to seven days or until delirium and agitation resolve. Rescue sedation may be provided with intravenous midazolam and fentanyl as clinically indicated. Delirium and agitation will be assessed regularly using validated tools such as the Confusion Assessment Method for the Intensive Care Unit and the Richmond Agitation-Sedation Scale.
  Arms: Dexmedetomidine Group

SUMMARY:
Traumatic brain injury is a serious and common medical condition that often requires admission to the intensive care unit and the use of mechanical ventilation. One of the most frequent and challenging complications in these patients is the development of delirium and agitation. These symptoms can prolong hospitalization, increase the risk of further brain injury, and complicate the medical and nursing care of the patient.

This interventional clinical trial is designed to compare the effects of two medications-haloperidol and dexmedetomidine-on the management of delirium and agitation in patients with traumatic brain injury admitted to the intensive care unit. Haloperidol is a traditional antipsychotic medication that is commonly used to manage agitation, but it may cause undesirable side effects such as movement disorders and disturbances in heart rhythm. Dexmedetomidine is a medication that acts on specific receptors in the nervous system to produce sedation and reduce agitation, and it is believed to cause fewer side effects related to breathing and movement.

The study will include forty adult patients with confirmed traumatic brain injury. These patients will be randomly assigned to receive either haloperidol or dexmedetomidine according to standard dosing guidelines. The study will evaluate and compare the following outcomes in both treatment groups: the presence and severity of delirium, the level of agitation, the total number of days the patient requires mechanical ventilation, the length of stay in the intensive care unit, the need for additional sedative medications, and the occurrence of any harmful effects from the study drugs.

To measure these outcomes, patients will be monitored using standardized tools that assess consciousness, agitation levels, and the presence of confusion. Additional medical examinations and laboratory tests will be conducted to ensure patient safety and collect relevant clinical data.

This study will be carried out in accordance with the ethical guidelines outlined in the Declaration of Helsinki and will follow internationally accepted standards for research involving human participants. Approval has been granted by the appropriate medical ethics committee at the Faculty of Medicine, Benha University. Informed consent will be obtained from all patients or their legal representatives before participation. The purpose of this research is to provide scientific evidence that can help doctors choose the most appropriate and safe medication for managing delirium and agitation in patients with traumatic brain injury who are being treated in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Confirmed diagnosis of traumatic brain injury
* Admission to the intensive care unit
* Currently receiving mechanical ventilation
* Richmond Agitation-Sedation Scale score between -5 and +4
* At least 48 hours have passed since ICU admission

Exclusion Criteria:

* Pre-existing neurological or psychiatric disorders (e.g., schizophrenia, bipolar disorder)
* Known allergy or contraindication to haloperidol or dexmedetomidine
* Significant hepatic or renal dysfunction
* Pregnant or breastfeeding women
* History of prolonged QT interval or other cardiac arrhythmias
* Use of long-term antipsychotic or sedative medications before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delirium | Daily for 7 days following initiation of intervention
  Delirium will be assessed using the Confusion Assessment Method for the Intensive Care Unit. The presence or absence of delirium will be documented daily. The aim is to compare the incidence of delirium between patients receiving haloperidol and those receiving dexmedetomidine. Evaluations will be conducted by trained healthcare personnel blinded to the intervention group.
Severity of Agitation | Daily for 7 days following initiation of intervention
  Agitation will be measured using the Richmond Agitation-Sedation Scale. Scores will be recorded daily to evaluate the severity of agitation in both treatment groups. The objective is to compare the effectiveness of haloperidol and dexmedetomidine in reducing agitation severity.
  Richmond Agitation-Sedation Scale (RASS) The Richmond Agitation-Sedation Scale is a 10-point scale ranging from +4 (combative) to -5 (unarousable), used to assess agitation and sedation levels in critically ill patients. Scores of +1 to +4 indicate increasing agitation, 0 indicates alert and calm, and -1 to -5 indicate increasing sedation. It is widely used in intensive care settings to guide sedation and evaluate treatment response.

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation | Up to 14 days after intervention initiation or until extubation
  The total number of days that each patient remains on mechanical ventilation will be recorded. The aim is to assess whether treatment with dexmedetomidine or haloperidol is associated with shorter ventilator dependency.
Length of Stay in the Intensive Care Unit | Up to 14 days after intervention initiation or until discharge from ICU
  The number of days each patient spends in the intensive care unit will be recorded to evaluate the impact of the assigned intervention on intensive care unit stay duration.
Need for Rescue Sedation | Within 7 days following initiation of intervention
  The number of patients requiring additional sedation with intravenous midazolam and fentanyl will be documented. This measure will compare the adequacy of haloperidol and dexmedetomidine in controlling delirium and agitation without supplemental sedatives.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this study will be shared, including data on demographics, intervention allocation, outcome measures (such as delirium incidence, agitation scores, ICU stay, and adverse events), and baseline clinical characteristics.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The individual participant data and supporting documents will be available beginning 6 months after publication of the primary results. The data will remain available for a period of 5 years.
Access Criteria: Qualified researchers affiliated with academic or medical institutions may request access to the de-identified data and supporting documents for the purpose of scientific research. Requests must be submitted to the principal investigator and will be evaluated based on scientific merit and alignment with the study's objectives. Approved researchers will sign a data access agreement and receive access via a secure data-sharing platform.